CLINICAL TRIAL: NCT05385796
Title: Study of Taping for Heel Fat Pad Syndrome (STEP): A Randomized Controlled Crossover Single-blind Clinical Trial
Brief Title: STEP Trial for Heel Fat Pad Syndrome
Acronym: STEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northwestern University (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Alison Chang, Associate Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: N-20210042
Record Dates: First submitted 2022-05-16; First posted 2022-05-23 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Heel Fat Pad Syndrome

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, participant-blinded trial, with a 2-arm crossover design.
Who Masked: Participant
Masking Description: To blind the participants, they will be told that both taping techniques have been used in the clinic and we want to investigate if they are effective and if one works better than the other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loop taping (Experimental): Loop taping of the heel fat pad
  Interventions: Other: Loop taping
- Control taping (Placebo Comparator): Control taping of the heel fat pad
  Interventions: Other: Control taping

INTERVENTIONS:
Other: Loop taping — The participant lays prone on the treatment table with his/her feet dangling off the table. The physiotherapist cleans the heel with alcohol wipes. Care is taken to avoid erasing skin markings for respective algometer and ultrasound assessment by these wipes. The therapist applies 1-inch-width Elastikon tape around the heel, encircling and bunching the fat pad to centralize it and enhance its fullness and resilience to compression. The tape starts at the middle distal end of the fat pad and loop around the periphery and ends by crossing the starting point at the middle distal end of the fat pad. Two to three overlapping loops will be applied to ensure strong support during weight-bearing activities. Participants will be instructed to wear the loop taping for 3 days and remove the taping after responding to an online survey 3-days post intervention.
  Arms: Loop taping
Other: Control taping — The participant lays prone on the treatment table with his/her feet dangling off the table. The physiotherapist cleans the heel with alcohol wipes. The therapist applies 1-inch-width Elastikon tape around the heel, lightly encircling the heel fat pad without any force/pressure or attempt to bunch or centralize the fat pad. The tape starts at the middle distal end of the fat pad and loop around the periphery and ends by crossing the starting point at the middle distal end of the fat pad. Two to three overlapping loops will be applied. Participants will be instructed to wear the control taping for 3 days and remove the taping after responding to an online survey 3-days post intervention.
  Arms: Control taping

SUMMARY:
The primary objectives of this study are to investigate the immediate and short-term effect of heel fat pad loop taping (experimental intervention) vs. control taping (control intervention) on pain and function in individuals with heel fat pad syndrome (HFPS). For mechanistic understanding of the effect of the loop taping, we will assess the immediate effect of taping on the pressure pain threshold and heel fat pad thickness.

DETAILED DESCRIPTION:
The study objectives are to investigate the immediate and short-term effect of heel fat pad loop taping (experimental intervention) vs. control taping (control intervention) on pain and function in individuals with heel fat pad syndrome (HFPS). We hypothesize that the fat pad loop taping is superior to control taping in immediate and short-term pain reduction and short-term function and mobility improvement. To understand potential mechanisms underlying the benefits of the looping taping, we will assess the immediate effect of taping on the pressure pain threshold and heel fat pad thickness. We hypothesize that applying fat pad loop taping will increase the pressure pain threshold (i.e., diminished pain sensitivity) recorded by a mechanical pressure algometer and increase fat pad thickness quantified by ultrasound. Despite being the second leading cause of plantar heel pain, RCTs for conservative management do not exist. Findings of this proposed project will provide much-needed evidence on effective non-pharmacological managements of HFPS.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 to 79 years of age
* History of plantar heel pain in either foot for at least one week and less than 3 years before enrollment
* Tenderness on palpation of the heel fat pad
* Self-reported worst unilateral or bilateral central heel pain of ≥ 3 on a 0-10 Numeric Pain Rating Scale (NPRS) during the past week
* Pain ≥ 3 on NPRS during at least one of two pain-aggravating activities of 30-sec static single leg standing OR barefoot 20-meter walking assessed during the enrollment screening and before the tape application

Exclusion Criteria:

* Primary diagnoses of plantar heel pain (e.g., plantar fasciopathy, posterior tibialis tendinopathy, or tarsal tunnel syndrome) other than HFPS
* Ultrasound-measured plantar fascia thickness ≥ 4mm, combined with clinical presentations of plantar fasciopathy
* BMI ≥ 35
* Systemic inflammatory arthritis
* Diabetes
* Lumbar radiculopathy
* Neurological conditions affecting gait and mobility
* Having received taping for HFPS within the last month
* Prior heel surgery

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Change from pre-intervention to immediately post-intervention in Numeric Pain Rating Scale (NPRS) during the most pain-aggravating activity | pre-intervention, immediately post-intervention
  The primary outcome is pain experienced during the most pain-aggravating activity (e.g., 30-sec static single leg standing or 20-meter barefoot walking) reported during the initial visit. Participants verbally select a value that corresponds with the intensity of pain that they experience. "0" means "no pain" and "10" means "pain as bad as you can imagine" or "worst pain imaginable". The NPRS, an 11-point (i.e., 0-10) measure of pain intensity, is recommended as a core outcome measure in clinical trials of chronic pain treatments and has excellent reliability and validity for adults with chronic musculoskeletal pain.

SECONDARY OUTCOMES:
Change from pre-intervention to 3 days post-intervention in Numeric Pain Rating Scale (NPRS) in the past 24 hours | pre-intervention, 3 days post-intervention
  Participants verbally select a value that corresponds with the average intensity of pain that they experience in the past 24 hours. Participants verbally select a value that corresponds with the intensity of pain that they experience. "0" means "no pain" and "10" means "pain as bad as you can imagine" or "worst pain imaginable". The NPRS, an 11-point (i.e., 0-10) measure of pain intensity, is recommended as a core outcome measure in clinical trials of chronic pain treatments and has excellent reliability and validity for adults with chronic musculoskeletal pain.
Change from pre-intervention to 3 days post-intervention in Foot Health Status Questionnaire (FHSQ) | pre-intervention, 3 days post-intervention
  The FHSQ is a self-administered questionnaire consisting of 13 items in 4 domains of foot pain (4 items), foot function (4 items), footwear (3 items), and general foot health (2 items). Each item is rated on a 5-point Likert scale from no (score =1) to severe (score = 5) pain, problems, or limitations. Responses to footwear questions are on a 5-point bipolar Likert scale from strongly disagree to strongly agree regarding shoe fit, discomfort wearing shoes, and shoewear available. Each domain score ranges from 0 (worst foot health) to 100 (optimal foot health). Higher scores indicate better foot health and quality of life. A validated Danish version of FHSQ is available. Good FHSQ test/retest and interrater/intrarater reliability and validity have been established for patients with foot disorders.
Global Rating of Change (GROC) | 3 days post-intervention
  Another core outcome measure for chronic musculoskeletal pain is the GROC, a widely used single-item instrument that asks each participant to indicate whether and to what extent they perceive change has occurred pre vs. post-intervention. This global rating is unique because, unlike other self-reported outcomes, it allows each participant to decide what he/she considers most important and relevant change. In the proposed study, participants will be queried "With respect to your heel pain, how would you describe it after the intervention compared to before the intervention?" and quantify the perceived change on a 7-point visual analogue scale of -3 to +3, where "-3" indicates "much worse", "0" indicates "no change", and "+3" indicates "much improved". GROC has been demonstrated to be a reliable and valid tool for musculoskeletal conditions.
Change from pre-intervention to immediately post-intervention in Pain sensitivity by pressure pain thresholds | pre-intervention, immediately post-intervention
  Pain sensitivity is quantified by measuring pressure pain thresholds (PPT) on the most painful spot on the heel fat pad, confirmed by palpation. Participants lay prone on the examination table, with the feet hanging freely over the edge of the table. The examiner places the 1-cm2 probe of a hand held mechanical pressure algometer perpendicular to the skin, and gradually increase the pressure at a rate of 30 kPa/s. Participants will report when the sensation changes from pressure, to the first onset of pain. This will be repeated three times, with a 30-second break between tests, and the average used for the analysis. The probe location will be marked on the skin to ensure placement consistency between pre- and post-intervention testing. The interrter and intrarater reliability of PPT assessment for patients with plantar heel pain was good at ICC 0.80-0.94 for intrarater and 0.75-0.92 for interrater.
Change from pre-intervention to immediately post-intervention in Heel fat pad thickness | pre-intervention, immediately post-intervention
  An ultrasound unit with a 6-13 MHz transducer frequency will be used to measure the heel fat pad thickness. Participants lay prone on the examination table, with the feet hanging freely over the edge of the table. The plantar fat pad will be marked by a sagittal midline; the ultrasound transducer will be placed on the midline for a transverse scan to measure the largest distance between the calcaneus and the skin. The average of two sonographic measurements will be used for analysis. The intrarater and interrater sonographic assessment of heel fat pad thickness was excellent with the intraclass correlation coefficients (ICCs) ranging from 0.81 to 0.96.

CONTACTS AND LOCATIONS:
Overall Officials: Alison H Chang, Principal Investigator — Northwestern University & Aalborg University
Locations (1):
- Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No